CLINICAL TRIAL: NCT04244591
Title: Glucocorticoid Therapy for Critically Ill Patients With Severe Acute Respiratory Infections Caused by COVID-19: a Prospective, Randomized Controlled Trial
Brief Title: Glucocorticoid Therapy for COVID-19 Critically Ill Patients With Severe Acute Respiratory Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Zhongda Hospital (Other); Zhongnan Hospital (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Glucocorticoid COVID-19
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-02

CONDITIONS: COVID-19 Infections
MeSH Terms: interventions — Steroids; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Placebo Comparator): standard care
  Interventions: Other: Standard care
- standard care + methylprednisolone therapy (Experimental): Methylprednisolone 40 mg q12h for 5 days
  Interventions: Drug: methylprednisolone therapy

INTERVENTIONS:
Drug: methylprednisolone therapy — Methylprednisolone 40 mg q12h for 5 days
  Other Names: Steroids
  Arms: standard care + methylprednisolone therapy
Other: Standard care — Standard care
  Arms: standard care

SUMMARY:
In this multi-center, randomized, control study, the investigators will evaluate the efficacy and safety of glucocorticoid in combination with standard care for COVID-19 patents with Severe acute respiratory failure.

DETAILED DESCRIPTION:
COVID-19 is a novel coronavirus that was initially outbreak in Wuhan, China. Severe acute respiratory infection with COVID-19 causes severe acute respiratory failure with substantial mortality. Currently, the standard care is supportive care, and no treatment is proven to be effective for this condition.

Glucocorticoid therapy is widely used among critically ill patients with other coronavirus infection such as SARS (severe acute respiratory syndrome) and MERS (Middle East respiratory syndrome). However, whether glucocorticoid improved the outcome of COVID-19 remains unknown. We hypothesized that glucocorticoid would improve the prognosis of patietns with COVID-19.

In this study, critically ill patients with COVID-19 were enrolled and randomized to receive ether standard care or standard care in combination with methylprednisolone therapy. The primary outcome is the difference of Murray lung injury score between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* PCR confirmed COVID-19 infection
* Symptoms developed more than 7 days
* PaO2/FiO2 < 200 mmHg
* Positive pressure ventilation (non-invasive or invasive) or high flow nasal cannula (HFNC) higher than 45 L/min for less than 48 hours
* Requiring ICU admission

Exclusion Criteria:

* pregnancy;
* patients currently taking corticosteroids (cumulative 400 mg prednisone or equivalent);
* Severe underlying disease, i.e. end stage of malignancy disease or end stage of pulmonary disease;
* Severe adverse events before ICU admission, i.e. cardiac arrest;
* Underlying disease requiring corticosteroids;
* Contraindication for corticosteroids;
* Recruited in other clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Lower Murray lung injury score | 7 days after randomization
  Murray lung injury score decreased more than one point means better outcome.The Murray scoring system range from 0 to 4 according to the severity of the condition.
Lower Murray lung injury score | 14 days after randomization
  Murray lung injury score decreased more than one point means better outcome.The Murray scoring system range from 0 to 4 according to the severity of the condition.

SECONDARY OUTCOMES:
The difference of PaO2/FiO2 between two groups | 7 days after randomization
  PaO2/FiO2 denotes ratio of arterial partial pressure of O2 and the fraction of inspired oxygen, with a higher PaO2/FiO2 means favorable outcome.
Lower Sequential Organ Failure Assessment (SOFA) score | 7 days after randomization
  Lower SOFA score means better outcome. The SOFA score system range from 0 to 24 according to the severity of the condition.
Mechanical ventilation support | 7 days after randomization
  Percentage of patients requiring Mechanical ventilation support
The difference of PaO2/FiO2 between two groups | 14 days after randomization
  PaO2/FiO2 denotes ratio of arterial partial pressure of O2 and the fraction of inspired oxygen, with a higher PaO2/FiO2 means favorable outcome.
Lower Sequential Organ Failure Assessment (SOFA) score | 14 days after randomization
  Lower SOFA score means better outcome. The SOFA score system range from 0 to 24 according to the severity of the condition.
Mechanical ventilation support | 14 days after randomization
  Percentage of patients requiring Mechanical ventilation support
Clearance of noval coronavirus | 14 days after randomization
  Clearance of noval coronavirus in upper respiratory tract or lower respiratory tract
All-cause mortality | 30 days after randomization
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Medical ICU,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arabi YM, Mandourah Y, Al-Hameed F, Sindi AA, Almekhlafi GA, Hussein MA, Jose J, Pinto R, Al-Omari A, Kharaba A, Almotairi A, Al Khatib K, Alraddadi B, Shalhoub S, Abdulmomen A, Qushmaq I, Mady A, Solaiman O, Al-Aithan AM, Al-Raddadi R, Ragab A, Balkhy HH, Al Harthy A, Deeb AM, Al Mutairi H, Al-Dawood A, Merson L, Hayden FG, Fowler RA; Saudi Critical Care Trial Group. Corticosteroid Therapy for Critically Ill Patients with Middle East Respiratory Syndrome. Am J Respir Crit Care Med. 2018 Mar 15;197(6):757-767. doi: 10.1164/rccm.201706-1172OC. PMID 29161116
- [Background] Auyeung TW, Lee JS, Lai WK, Choi CH, Lee HK, Lee JS, Li PC, Lok KH, Ng YY, Wong WM, Yeung YM. The use of corticosteroid as treatment in SARS was associated with adverse outcomes: a retrospective cohort study. J Infect. 2005 Aug;51(2):98-102. doi: 10.1016/j.jinf.2004.09.008. PMID 16038758
- [Background] Raghavendran K, Napolitano LM. Definition of ALI/ARDS. Crit Care Clin. 2011 Jul;27(3):429-37. doi: 10.1016/j.ccc.2011.05.006. PMID 21742209
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091